CLINICAL TRIAL: NCT02458703
Title: Hypoxemia, Dyspnea, and Exercise Tolerance in Patients With Pulmonary Arteriovenous Malformations , With and Without Airflow Obstruction
Brief Title: Cardiopulmonary Exercise Testing to Evaluate Pulmonary AVMs With and Without Airflow Obstruction
Acronym: ExercisePAVM2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CLS 2015/1; 15/LO/0598 (Other: National Research Ethics Service, UK)
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-04

CONDITIONS: Pulmonary Arteriovenous Malformations; Hereditary Hemorrhagic Telangiectasia; Asthma; COPD
Keywords: workload; oxygen level; oxygen consumption; breathing reserve; ventilatory efficiency
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test; Clostridium perfringens epsilon-toxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with pulmonary AVMs and no airflow obstruction (Experimental): 30 patients with pulmonary AVMs and no airflow obstruction will undergo cardiopulmonary exercise testing
  Interventions: Other: Cardiopulmonary exercise test
- Patients with pulmonary AVMs and airflow obstruction (Experimental): 30 patients with pulmonary AVMs and airflow obstruction will undergo cardiopulmonary exercise testing
  Interventions: Other: Cardiopulmonary exercise test

INTERVENTIONS:
Other: Cardiopulmonary exercise test — Subjects will have the test in the Exercise Suite of Hammersmith Hospital, London, UK. They will have painless skin probes placed on their fingers, chest, and legs to monitor heart rate, ECG, blood oxygen levels, and oxygen delivery during the test. Subjects will also be shown how to breathe through a mouthpiece with a nose clip on, and how to indicate on a sliding device whether they feel breathless. They will then start cycling against a very low resistance at a steady speed. As long as they feel comfortable, there will be a gradual increase in work load until they feel they cannot keep going at the same speed. They can also stop sooner for any reason. Afterwards, while they are "cooling down", they will fill in a short questionnaire describing how they feel. 20-30mls of blood will be taken for analysis.
  Other Names: CPET

SUMMARY:
Pulmonary arteriovenous malformations (PAVMs) are a rare vascular condition affecting the lungs. PAVMs lead to low blood oxygen levels, yet are very well tolerated by patients. This study will examine the exercise capacity of PAVM patients using formal cardiopulmonary exercise tests performed on a stationary bicycle, and whether this is affected by the presence of concurrent airflow obstruction, such as due to asthma.

DETAILED DESCRIPTION:
It is well known that the lung is the site at which oxygen enters the blood stream, diffusing from the alveolar air sacs into the pulmonary capillaries. This newly oxygenated blood is carried to the heart in the pulmonary veins, then passes into the systemic circulation to provide oxygen to the tissues.

Patients with pulmonary arteriovenous malformations (PAVMs) have abnormal vascular connections between pulmonary arteries and pulmonary veins in the lung. Blood flowing through PAVMs therefore bypasses the oxygenation sites in the pulmonary capillaries. Low blood oxygen levels (hypoxemia) is frequent in PAVM patients but breathlessness (dyspnea) is not. The investigators have shown that dyspnea was not a common presenting complaint in a large UK series, and that there is little correlation between severity of dyspnea in PAVM patients, and blood oxygen levels.

In this study the investigators will address the question "Do PAVM patients have lower exercise tolerance if they have concurrent airflow obstruction?" The primary outcome measure will be the total body oxygen consumption in mls/min/kg, at peak exercise (the V[dot]O2 peak (also known as "VO2 max")).

The investigators will address this by first performing standardised cardiopulmonary exercise testing, as used in the clinic and our previous study (11/H0803/9), on age and sex matched patients with PAVMs. 30 will be recruited with airflow obstruction, and 30 without airflow obstruction. Physiological parameters will be compared, to test the null hypothesis that the impact of exercise on PAVM patients' cardiopulmonary systems does not differ according to the presence or absence of airflow obstruction. Cellular and molecular methods will be used to dissect mechanistic pathways.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Pulmonary AVMs no airflow obstruction: Pulmonary AVMs confirmed by CT scan and no evidence or history of airflow obstruction on clinical grounds, or by spirometric evaluations.
* Pulmonary AVMs with airflow obstruction: Pulmonary AVMs confirmed by CT scan and evidence or history of airflow obstruction on clinical grounds, and/or by spirometric evaluations (such as FEV1/VC ratio <80%).

Exclusion Criteria:

* Inability to provide informed consent
* Any known cardiovascular abnormality including a history of syncope (faintness, dizziness, lightheadedness or loss of consciousness due to an abnormality of the cardiovascular system).
* Current respiratory tract infection (eg a cold).
* Pregnancy.
* Claustrophobia or needle phobia

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Total body oxygen consumption in mls/min/kg, at peak exercise (VO2 max). | Same day (within 1 hour), at end of exercise study
  Of the many measurements and derived indices that can be measured during cardiopulmonary exercise testing, the peak consumption of oxygen (VO2 max) is perhaps the best indicator of integrated cardiorespiratory capacity. The principle research question will therefore test the null hypothesis that "The VO2 max does not differ between PAVM patients with and without airflow obstruction."

SECONDARY OUTCOMES:
Breathing reserve | Same day (within 1 hour), at end of exercise study
  We will also test in univariate and multiple regression analyses whether breathing reserve differs between PAVM patients with and without airflow obstruction.
Ventilatory efficiency | Same day (within 1 hour), at end of exercise study
  We will also test in univariate and multiple regression analyses whether ventilatory efficiency differs between PAVM patients with and without airflow obstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, PhD FRCP, Principal Investigator — Hammersmith Hospital, Du Cane Rd, London, United Kingdom, W12 0NN

REFERENCES:
- [Background] Howard LSGE, Santhirapala V, Murphy K, Mukherjee B, Busbridge M, Tighe HC, Jackson JE, Hughes JMB, Shovlin CL. Cardiopulmonary exercise testing demonstrates maintenance of exercise capacity in patients with hypoxemia and pulmonary arteriovenous malformations. Chest. 2014 Sep;146(3):709-718. doi: 10.1378/chest.13-2988. PMID 24676541